CLINICAL TRIAL: NCT01990157
Title: Safety, Tolerability, Pharmacodynamics and Efficacy Study of TAB08 in Patients With Rheumatoid Arthritis in Which Methotrexate (MTX) Treatment is Not Effective
Brief Title: Safety, Tolerability, Pharmacodynamics and Efficacy Study of TAB08 in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Theramab LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAB08_RA01
Record Dates: First submitted 2013-11-05; First posted 2013-11-21 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — TGN-1412

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAB08 (Experimental): Multiple TAB08 administrations as intravenous infusions.
  Interventions: Drug: TAB08

INTERVENTIONS:
Drug: TAB08 — Weekly intravenous administration in escalating doses.
  Other Names: Theralizumab

SUMMARY:
This study is in two stages:

Stage 1 purpose is to assess safety, tolerability, and efficacy of multiple TAB08 doses in patients with active Rheumatoid Arthritis in which methotrexate (MTX) treatment is not enough effective.

Stage 2 purpose is to assess efficacy parameters (ACR criteria) of at least one selected TAB08 dose in extended patient population with active Rheumatoid Arthritis in which methotrexate (MTX) treatment with at least 10 mg/week is not enough effective.

DETAILED DESCRIPTION:
Stage 1 is designed as standard phase 1 study with one arm and sequential dose cohorts with ascending doses. Each patient in each dose cohort will be administered TAB08 several times. After last TAB08 administration each patient will undergo investigational-treatment-free follow-up period.

At Stage 2 at least one TAB08 dose, selected during Stage 1 will be studied during longer timeframe in extended patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must sign and date informed consent prior to any study procedures.
2. Male and female patients aged 18-65 years.
3. Rheumatoid arthritis (RA) diagnosed from 6 months to 10 years ago in accordance with American College of Rheumatology (ACR) diagnostic criteria of rheumatoid arthritis, 1987, or ACR / European League against Rheumatism (EULAR), 2010.
4. Patients for whom standard treatment does not result in sufficient control of symptoms of RA, per investigator opinion.
5. Treatment with Methotrexate for at least 3 months before Screening visit, and a stable dose of ≥ 10 mg weekly for at least 28 days before the first infusion of the study drug. Patients should be also treated with folic acid.
6. Active disease of RA despite standard treatment:

   1. At least 6 out of 66 joints are swollen and at least 6 out of 68 joints are painful.
   2. Level of C-reactive protein >= 15 mg/L or erythrocyte sedimentation rate >= 28 mm/hour or morning stiffness > 45 minutes.
7. Rheumatoid factor > 20 IU/mL.
8. Adequate hematological, renal and hepatic laboratory values.
9. For men and women of childbearing potential: consent to use double barrier methods of contraception during the entire study period.

Exclusion Criteria:

1. Use of other disease-modifying antirheumatic drugs (DMARDs) except for Methotrexate within 4 weeks before the treatment initiation. Use of Leflunomide within 8 weeks before the first study drug infusion. Use of biological immunosuppressive drugs (Adalimumab, Etanercept, Infliximab, Anakinra, Abatacept and others) 2 months before the first study drug administration. Use of Rituximab within 12 months before the first study drug administration.
2. Change of Methotrexate dose within 4 weeks before study treatment initiation.
3. Any autoimmune disease except for rheumatoid arthritis and dry keratoconjunctivitis.
4. Functional grade IV based on American College of Rheumatology scale.
5. Active rheumatoid vasculitis.
6. Any systemic diseases related to joint inflammation.
7. Pregnant and breastfeeding women.
8. Women with childbearing potential refusing to use effective contraceptive methods during the entire study period.
9. Any active infectious disease or tuberculosis at the moment or within 2 weeks before inclusion into the study.
10. Syphilis, hepatitis В, С, HIV-infection or tuberculosis based on the results of laboratory tests at Screening visit.
11. Vaccination with live or attenuated vaccines within 6 weeks before the first study drug administration; planned vaccination during the study period.
12. Medical history of recurrent clinically significant infections.
13. Primary or secondary immunodeficiency.
14. Medical history of malignant oncologic diseases except for excised basal cell skin cancer.
15. Treatment with glucocorticosteroids (GKS) in a dose corresponding to over 12.5 mg/day of prednisolone equivalent, or change of GKS dose as well as treatment with intraarticular, i/m or i/v injections of GKS within 4 weeks before the first infusion of the study drug except for topical low active GKS, GKS in eardrops or eyedrops/ointment, inhalant GKS in a stable dose for the entire study period.
16. Dose change of non-steroid anti-inflammatory agents within 4 weeks before first infusion of the study drug.
17. Any factors that per investigator opinion might prevent patient from adhering to the visit schedule or performing study requirements.
18. Participation in any other clinical study of an experimental drug within 3 months or within 5 elimination half-lives (depending on whichever is longer) before the first infusion of the study drug.
19. Medical history of the following diseases: myocardial infarction, angina pectoris, bronchial asthma, chronic obstructive pulmonary disease or other cardiovascular or respiratory pathology which is considered serious by investigator.
20. Current uncontrolled pathology of renal, endocrine, hematology or central nervous system.
21. Alcohol and/or drug abuse within 1 year before first study drug administration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity in every dose cohort | From study drug infusion (Day 1) untill week 2 (Day 15) for each patient

SECONDARY OUTCOMES:
Number of adverse events | From study drug infusion (Day 1) untill the end of study stage 1 (Day 85)

OTHER OUTCOMES:
Pharmacokinetics parameters of TAB08 after single and multiple i.v. administrations | From study drug infusion (Day 1) untill Week 4 (Day 29)
  Following specific pharmacokinetics parameters will be used:
  C max - maximal concentration, AUC(0-t) - area under the curve concentration-time until the last time point of concentration measurement, AUC(0-∞) - area under the curve concentration-time extrapolated to infinity, T1/2 - final elimination half-life, Lambda z - elimination rate constant, CL - clearance, Vss - volume of distribution in steady state, C trough - trough concentration after multiple administration.
Proportion of patients with American College of Rheumatology (ACR) 20 (50, 70) response criteria after 4 weeks of TAB08 treatment | From study drug infusion (Day 1) untill the Week 4 (Day 29)
Proportion of patients with ACR20 (50, 70) response criteria after 4 weeks of TAB08 treatment at the end of study stage 1 | From study drug infusion (Day 1) untill tenf of study stage 1 (Day 85)

CONTACTS AND LOCATIONS:
Overall Officials: Daniil G Nemenov, M.D., Study Director — Theramab LLC
Locations (2):
- Russia (2):
  - State Scientific and Research Rheumatology Institute, Moscow
  - Clinical Emergency Hospital of Yaroslavl, Yaroslavl